CLINICAL TRIAL: NCT06124027
Title: What is the Effect of Deep Procedural Sedation With HFNOT on the tcPCO2, mitoPO2 and mitoVO2.
Brief Title: Impact of Sedation With HFNOT on tcPCO2, mitoPO2 and mitoVO2.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Calvin de Wijs, MSc (Other)
Responsible Party: Sponsor-Investigator, Calvin de Wijs, MSc, M.D., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-2022-0421; NL81086.078.22 (Other: The Central Committee on Research Involving Human Subjects.)
Record Dates: First submitted 2023-10-31; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Sedation Complication; High Flow Nasal Oxygen Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Monitoring tcPCO2 and mitoPO2 — Monitoring tcPCO2 using SenTec and mitoPO2 using COMET

SUMMARY:
Deep procedural sedation has seen an increased use indication over the last couple of years aided by the introduction of high flow nasal oxygen therapy (HFNOT) during these procedures. However, this level of deep sedation does come with the increased risk of examining whether a patient is adequately ventilated during this procedure.

The definition of deep sedation is: 'a drug-induced depression of consciousness during which patients cannot be easily aroused but respond purposefully following repeated or painful stimulation. The ability to independently maintain ventilatory function may be impaired. Patients may require assistance in maintaining a patent airway, and spontaneous ventilation may be inadequate. Cardiovascular function is usually maintained.' As the definition showed there may be an insufficient ventilation during deep sedation. Therefore, HFNOT is used to ensures that the peripheral oxygen saturation is sufficient. However, there are two potential disadvantages. HFNOT can mask the presence of an insufficient respiratory minute volume and an insufficient gas exchange, which can lead to high arterial CO2 (paCO2) levels. Another risk associated with HFNOT is the fact that high oxygen levels are toxic, and prolonged exposure to high partial oxygen pressures, can cause oxidative damage to cell membranes, collapse of the alveoli in the lungs, retinal detachment, and seizures. Most of this damage can be explained by hyperoxia that increases the 'leak' of electrons from the mitochondrial electron transport chain and the resulting increased generation of reactive oxygen species (ROS). Low paCO2 levels and hyperoxia cannot be examined using standard monitoring techniques therefore, this study will use the transcutaneous carbon dioxide (tcPCO2) a proven technique which correlates well to the arterial CO2 (paCO2) to evaluate whether there is an adequate level of ventilation during deep procedural anesthesia with HFNOT. Moreover, the cutaneous mitochondrial oxygenation (mitoPO2) will be monitored to determine the effects that deep procedural sedation with HFNOT has on the cellular oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Acceptable proficiency of the Dutch language
* Scheduled for a procedure requiring deep procedural sedation with HFNOT.

Exclusion Criteria:

* Porphyria
* Known intolerance to components of the ALA plaster
* Presence of mitochondrial disease
* Pregnancy/lactation
* Patients with skin lesions on the measurement location which impede measurements
* Incapability to provide inform consent, due to a mental condition interfering with the ability to understand the provided information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of patients undergoing procedures which require deep procedural sedation with HFNOT.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
tcPCO2. | up to 6 hours
  To examine the effects of deep procedural sedation and use of HFNOT on the tcPCO2.
mitoPO2 | up to 6 hours
  To determine the effects of deep procedural sedation and use of HFNOT on the mitoPO2

SECONDARY OUTCOMES:
mitoVO2 | up to 6 hours
  To determine the effects of deep procedural sedation and use of HFNOT on the mitoVO2

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided